CLINICAL TRIAL: NCT02953691
Title: Exploring the Impact of Perioperative Galacto-Oligosaccharides (GOS) on Stress, Anxiety and Cognition
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Study Substance
Sponsor: Jeff Taekman, M.D. (Other)
Responsible Party: Sponsor-Investigator, Jeff Taekman, M.D., Professor of Anesthesiology, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00075000
Record Dates: First submitted 2016-10-24; First posted 2016-11-03 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Anxiety; Pain; Surgery
Keywords: perioperative; surgery; pain; anxiety; post operative cognitive dysfunction; cognition
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — 4'-galactooligosaccharide; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Galacto-Oligosaccharides (GOS) (Experimental): Clasado Biosciences Limited will provide Bimuno Pastilles for the clinical trial. Each pastille contains 0.92g GOS and will be taken 3 times per day. Following informed consent, subjects will be issued prepackaged GOS pastilles to be taken three times daily up until the evening prior to surgery. Subjects will be randomly assigned to receive GOS prebiotics. Each subject has an equal chance of receiving GOS or placebo. GOSn will be administered in the hospital when patient reinstitutes oral intake. GOS will be issued to each subject to last until the day of their scheduled follow-up for POCD (approximately 1.5 months post surgery).
  Interventions: Drug: Galacto-Oligosaccharide
- Maltodextrin (Placebo) (Placebo Comparator): Clasado Biosciences Limited will provide placebo (Maltodextrin) for the clinical trial. Each pastille contains maltodextrin and will be taken 3 times per day. Following informed consent, subjects will be issued prepackaged pastilles to be taken three times daily up until the evening prior to surgery. Subjects will be randomly assigned to receive GOS prebiotics or placebo. Each subject has an equal chance of receiving GOS or placebo. Placebo will be administered in the hospital when patient reinstitutes oral intake. Placebo will be issued to each subject to last until the day of their scheduled follow-up for POCD (approximately 1.5 months post surgery).
  Interventions: Drug: Maltodextrin (Placebo)

INTERVENTIONS:
Drug: Galacto-Oligosaccharide — Mixture produced from lactose utilizing the transgalactosidic activity of Bifidobacterium bifidum NCIMB 41171 beta-galactosidase
  Arms: Galacto-Oligosaccharides (GOS)
Drug: Maltodextrin (Placebo) — Maltodextrin is a polysaccharide commonly used as a food additive. It is produced from starch by partial hydrolysis.
  Arms: Maltodextrin (Placebo)

SUMMARY:
The overall objective of this proposal is to explore the association between the administration of the prebiotics GOS (trade name: Bimuno Travelaid; generic name:B galacto-oligosaccharides) with pain, anxiety, and cognitive function in the perioperative period. The investigators' central hypothesis is subjects who consume GOS in the perioperative period will demonstrate lower levels of salivary cortisol before, during, and after their operative procedures. In addition, the investigators expect subjects who consume GOS to have lower perceived levels of anxiety during the perioperative period. Finally, the investigators hypothesize that subjects who consume perioperative GOS will perform better on tests of cognition in the postoperative period. Such a finding would be beneficial in that administration of GOS in the perioperative period offers a safe and inexpensive adjunct to current medical management of perioperative anxiety.

DETAILED DESCRIPTION:
AIM 1: In anterior cervical decompression and fusion (ACDF) subjects, explore the association between prebiotics, anxiety, and pain.

Studies have recently elucidated a link between certain prebiotics and lower perceived anxiety as well as biomarkers of stress. In this aim the investigators will explore the association between consumption of prebiotics and their relationship to perioperative anxiety / physiological stress response. The investigators hypothesize that subjects who receive prebiotics will have lower perioperative anxiety and stress versus control as measured by standardized surveys and biomarkers. Furthermore, the investigators hypothesize that lower anxiety will result in lower postoperative pain scores.

AIM 2: In ACDF patients, explore the association between GOS and post-operative cognitive dysfunction.

Stress and anxiety is known to impair cognitive function. In addition, in preclinical studies, the administration of distinct keystone bacterial strains improves cognitive function in an anxious mouse model. In humans, prebiotics and probiotics have been shown to ameliorate the stress response. In this aim the investigators seek to explore the association between prebiotics and perioperative cognitive outcomes in humans. The investigators will perform cognitive function testing using the same time-tested battery used in the department to study post-operative cognitive decline (POCD). Subjects will be tested for cognitive function preoperatively (T1) and at 1.5 months post-op (T4). The investigators hypothesize that patients receiving prebiotics during the perioperative period will show less post-operative cognitive dysfunction than controls.

A total of 8 subjects will be recruited from the Neurosurgery Clinics of Duke University Health System. The target population will include subjects undergoing ACDF. Exclusion criteria will include: pregnant women, age<21 years, a diagnosis of depression, mental or behavioral disorder, recent anxiolytic use, long-term opiate use, oral contraceptive use, or recent antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing anterior cervical discectomy and fusion

Exclusion Criteria:

* Pregnancy
* Breast Feeding Women
* Diagnosis of Depression
* Diagnosis of mental or behavioral disorder
* Recent anxiolytic use (within 1 week of enrollment)
* Long-term opiate use (greater than 1 week prior to enrollment)
* Recent systemic steroid use (within 1 week of enrollment)
* Diagnosis of cancer
* Oral or intravenous antibiotic use within 1 month of enrollment

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Waking Salivary Cortisol | Morning after Preop Clinic Visit (2 weeks prior to surgery), 2-hours before surgery, 1-day after surgery, 6-week follow-up visit

SECONDARY OUTCOMES:
Changes in pain perception | Preop Clinic Visit (2 weeks prior to surgery), 2-hours before surgery, 30 minutes after surgery, 1-day after surgery, 6 week follow-up visit
  Collected through Visual Analog Scale.
Changes in cognition | Preop Clinic Visit (2 weeks prior to surgery), 6 week follow-up visit
  Hopkins Verbal Learning Test - Revised (HVLT-R)
Changes in perceived stress | Preop Clinic Visit (2 weeks prior to surgery), 2-hours before surgery, 1-day after surgery, 6 week follow-up visit
  Subjects will complete web-based versions of the State-Trait Anxiety Scale.
Changes in perceived stress | Preop Clinic Visit (2 weeks prior to surgery), 2-hours before surgery, 1-day after surgery, 6 week follow-up visit
  Subjects will complete web-based versions Hospital Anxiety and Depression Scale-HADS.
Changes in perceived stress | Preop Clinic Visit (2 weeks prior to surgery), 2-hours before surgery, 30 minutes after surgery, 1-day after surgery, 6 week follow-up visit
  Subjects will complete web-based versions Visual Analog Anxiety Scale.
Changes in cognition | Preop Clinic Visit (2 weeks prior to surgery), 6 week follow-up visit
  Randt Short Story Memory Test
Changes in cognition | Preop Clinic Visit (2 weeks prior to surgery), 6 week follow-up visit
  Modified Visual Reproduction Test from the Wechsler Memory Scale
Changes in cognition | Preop Clinic Visit (2 weeks prior to surgery), 6 week follow-up visit
  Weschsler Adult Intelligence Scale - Revised (WAIS-R)
Changes in cognition | Preop Clinic Visit (2 weeks prior to surgery), 6 week follow-up visit
  Trail Making Test
Changes in cognition | Preop Clinic Visit (2 weeks prior to surgery), 6 week follow-up visit
  Grooved Pegboard
Changes in cognition | Preop Clinic Visit (2 weeks prior to surgery), 6 week follow-up visit
  Mini Mental Status Exam (MMSE)
Suicidal ideation and behavior | Preop Clinic Visit (2 weeks prior to surgery), 2-hours before surgery, 1-day after surgery, 6 week follow-up visit
  Columbia-Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Taekman, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt K, Cowen PJ, Harmer CJ, Tzortzis G, Errington S, Burnet PW. Prebiotic intake reduces the waking cortisol response and alters emotional bias in healthy volunteers. Psychopharmacology (Berl). 2015 May;232(10):1793-801. doi: 10.1007/s00213-014-3810-0. Epub 2014 Dec 3. PMID 25449699
- [Background] Tillisch K. The effects of gut microbiota on CNS function in humans. Gut Microbes. 2014 May-Jun;5(3):404-10. doi: 10.4161/gmic.29232. Epub 2014 May 16. PMID 24838095